CLINICAL TRIAL: NCT05365217
Title: A Multi-centre, Open-label Trial Evaluating Efficacy, Safety and Pharmacokinetics of Nonacog Beta Pegol When Used for Treatment and Prophylaxis of Bleeding Episodes in Chinese Patients With Haemophilia B
Brief Title: A Research Study Investigating Nonacog Beta Pegol (N9-GP) for Treatment and Prevention of Bleedings in Chinese People With Haemophilia B
Acronym: Paradigm9
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN7999-4670; 2021-004947-25 (EudraCT Number); U1111-1260-0438 (Other: World Health Organization (WHO)); CTR20220763 (Registry Identifier: China Drug Trials (China))
Record Dates: First submitted 2022-05-04; First posted 2022-05-09 (Actual); Results first posted 2025-05-31 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Haemophilia B
MeSH Terms: conditions — Hemophilia B | interventions — nonacog beta pegol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Arm A - Nonacog beta pegol (On-demand/Prophylaxis) (Experimental): Participants on on-demand treatment for 28 weeks, thereafter prophylactic treatment
  Interventions: Drug: Nonacog beta pegol
- Arm B - Nonacog beta pegol (Prophylaxis) (Experimental): Participants on prophylactic treatment only
  Interventions: Drug: Nonacog beta pegol

INTERVENTIONS:
Drug: Nonacog beta pegol — Nonacog beta pegol is administered as intravenous injections. Participants will receive nonacog beta pegol as prophylaxis, as on-demand for treatment of bleeding episodes and in relation to surgery.

SUMMARY:
The study investigates how well the medicine called nonacog beta pegol (N9-GP) works in Chinese people with haemophilia B. Participants will be treated with N9-GP. This is a medicine that doctors can already prescribe in other countries. The medicine will be injected into a vein (intravenous injection). At the visits to the clinic, the medicine will be injected by the study doctor. When treating themselves at home, participants inject the medicine using a needle and vial set. The study will last for about 12-16 months. The participants will have between 9 and 19 visits to the clinic and possibly also some phone calls with the study doctor. At all visits to the clinic, the participants will have blood samples taken.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained before any trial-related activities. Trial-related activities are any procedures that are carried out as part of the trial, including activities to determine suitability for the trial.
* Male Chinese patient with moderate to severe congenital haemophilia B with a factor IX (FIX) activity less than or equal to 2 percent according to medical records.
* Aged 12-70 years (both inclusive) at the time of signing informed consent.
* History of at least 100 exposure days (EDs) to products containing FIX.1.
* Patients currently on prophylaxis or patients currently treated on-demand with at least 6 bleeding episodes during the last 12 months or at least 3 bleeding episodes during the last 6 months.
* The patient, legally authorised representative (LAR) and/or caregiver are capable of assessing a bleeding episode, keeping a diary, performing home treatment of bleeding episodes and otherwise following the trial procedures.

Exclusion Criteria:

* Known or suspected hypersensitivity to trial product or related products.
* Previous participation in this trial. Participation is defined as signed informed consent.
* Participation in any clinical trial of an approved or non-approved investigational medicinal product within 5 half-lives or 30 days from screening, whichever is longer.
* Known history of FIX inhibitors based on existing medical records, laboratory report reviews and patient and LAR interviews.
* Current FIX inhibitors greater than or equal to 0.6 Bethesda unit (BU).
* HIV positive, defined by medical records, with CD4+ count less than or equal 200 per microlitre (μL) and a viral load greater than 200 particles per microlitre or greater than 400000 copies per millilitre (mL) within 6 months of the trial entry. If the data are not available in the medical records within the last 6 months, then the test must be performed at the screening visit.
* Congenital or acquired coagulation disorder other than haemophilia B.
* Previous arterial thrombotic events (e.g. myocardial infarction and intracranial thrombosis) or previous deep venous thrombosis or pulmonary embolism (as defined by available medical records).
* Hepatic dysfunction defined as aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) greater than 3 times the upper limit of normal combined with total bilirubin greater than 1.5 times the upper limit of normal at screening.
* Renal impairment defined as estimated glomerular filtration rate (eGFR) less than or equal to 30 mL/min/1.73 m^2 for serum creatinine measured at screening.
* Any disorder, except for conditions associated with haemophilia B, which in the investigator's opinion might jeopardise the patient's safety or compliance with the protocol.
* Platelet count less than 50×10^9/L at screening.
* Immune modulating or chemotherapeutic medication.
* Mental incapacity, unwillingness or language barriers precluding adequate understanding or cooperation.

Ages: 12 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-05-18 (Actual); Primary Completion 2024-04-11 (Actual); Study Completion 2024-05-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency dept. 2834, Study Director — Novo Nordisk A/S
Locations (14):
- China (14):
  - Beijing Children's Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Fujian Medical University Union Hospital-Hematology, Fuzhou, Fujian
  - Nanfang Hospital, Southern Medical University-Haematology, Guangzhou, Guangdong
  - The Affiliated Hospital of Guizhou Medical University-Hematology, Guiyang, Guizhou
  - Henan Cancer Hospital-Hematology, Zhengzhou, Henan
  - Tongji Hospital, Tongji Medical College of HUST-Hematology, Wuhan, Hubei
  - Xiangya Hospital Central-South University, Changsha, Hunan
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - Jinan Central Hospital, Jinan, Shandong
  - The Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - Institute of Hematology and Blood Diseases Hospital, Tianjin-Hematology, Tianjin, Tianjin Municipality
  - The Second Affiliated Hospital of Kunming Medical University, Kunming, Yunnan
  - Children's Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This trial was conducted at 15 sites that enrolled participants in 1 country (China mainland).
Pre-assignment Details: A total of 30 participants were exposed to trial products, of which 15 participants were in Arm A (on demand/Prophylaxis) treatment group and 15 in Arm B (Prophylaxis) treatment group.
Groups:
- Arm A: Nonacog Beta Pegol (On-demand, Then Prophylaxis): Participants received intravenous injections of nonacog beta pegol (on-demand treatment for 28 weeks during treatment period 1, followed by 40 international unit per kilogram (IU/kg) for mild or moderate bleeds and 80 IU/kg for severe bleeds, with additional doses as needed if the initial treatment showed no effect during treatment period 2) until 30 exposure days (EDs) to nonacog beta pegol in the entire trial were fulfilled.
- Arm B: Nonacog Beta Pegol (Prophylaxis): Participants received intravenous injections of 40 IU/kg nonacog beta pegol once weekly (prophylactic treatment with nonacog beta pegol at a dose of 40 IU/kg weekly) until 50 EDs (including treatment of breakthrough bleeds) and 50 weeks in the entire trial were fulfilled.
Period: Treatment Period 1
Arm/Group | Arm A: Nonacog Beta Pegol (On-demand, Then Prophylaxis) | Arm B: Nonacog Beta Pegol (Prophylaxis)
Started | 15 | 15
Completed | 14 | 15
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Period: Treatment Period 2
Arm/Group | Arm A: Nonacog Beta Pegol (On-demand, Then Prophylaxis) | Arm B: Nonacog Beta Pegol (Prophylaxis)
Started | 14 | 15
Completed | 14 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Results were based on the FAS which included all participants exposed to N9-GP in this trial.
Groups:
- Arm A: Nonacog Beta Pegol (On-demand, Then Prophylaxis): Participants received intravenous injections of nonacog beta pegol (on-demand treatment for 28 weeks during treatment period 1, followed by 40 IU/kg for mild or moderate bleeds and 80 IU/kg for severe bleeds, with additional doses as needed if the initial treatment showed no effect during treatment period 2) until 30 exposure days (EDs) to nonacog beta pegol in the entire trial were fulfilled.
- Total: Total of all reporting groups
Arm/Group | Arm A: Nonacog Beta Pegol (On-demand, Then Prophylaxis) | Arm B: Nonacog Beta Pegol (Prophylaxis) | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Mean (Standard Deviation); unit: Years] | 29.9 (7.7) | 26.9 (9.7) | 28.4 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 15 | 15 | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 15 | 15 | 30
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 15 | 15 | 30
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Haemostatic Effect of Nonacog Beta Pegol When Used for Treatment of Bleeding Episodes During on Demand and Prophylaxis (PPX)
Description: Haemostatic effect of N9-GP for treatment of bleeding episodes was assessed by 4-point response scale: none, moderate, good or excellent. Evaluation during trial was done by participant and/or parent(s)/caregiver within approximately 8 hours after a single injection as follows: Excellent: Abrupt pain relief and/or clear improvement in objective signs of bleeding within approximately 8 hrs after a single injection; Good: Definite pain relief and/or improvement in signs of bleeding within approximately 8 hrs after a single injection, but possibly requiring more than one injection for complete resolution; Moderate: Probable or slight beneficial effect within approximately 8 hours after the first injection, but usually requiring more than one injection; None: No improvement, or worsening of symptoms.
Time Frame: From start of treatment (week 0) until end of treatment (up to week 50)
Population: Results were based on the FAS which included all participants exposed to N9-GP in this trial.
Measure: Number; unit: Bleeding Episodes
Units Other Than Participants: Bleeding Episodes
Groups:
- Arm A: Nonacog Beta Pegol (On-demand): Participants received intravenous injections of nonacog beta pegol on-demand treatment for 28 weeks.
- Arm A: Nonacog Beta Pegol (Prophylaxis): Participants received intravenous injections of nonacog beta pegol prophylactic treatment with 40 IU/kg for mild or moderate bleeds and 80 IU/kg for severe bleeds, with additional doses as needed if the initial treatment showed no effect, until 30 EDs to nonacog beta pegol in the entire trial were fulfilled.
Arm/Group | Arm A: Nonacog Beta Pegol (On-demand) | Arm A: Nonacog Beta Pegol (Prophylaxis) | Arm B: Nonacog Beta Pegol (Prophylaxis)
Number analyzed (Participants) | 15 | 14 | 15
Number analyzed (Bleeding Episodes) | 215 | 4 | 43
Bleeding Episodes
  Excellent | 203 | 3 | 26
  Good | 8 | 1 | 16
  Moderate | 3 | 0 | 1
  None | 1 | 0 | 0
  Missing | 0 | 0 | 0

2. Secondary Outcome: Number of Treated Bleeding Episodes During Prophylaxis (PPX) Treatment (Arm B Only)
Description: Number of bleeding episodes per year data is reported. Annualised bleeding rate (ABR) is the number of bleeding episodes per year.
Time Frame: From start of treatment (week 0) until end of treatment (week 50)
Population: Results were based on the FAS which included all participants exposed to N9-GP in this trial.
Measure: Median (Inter-Quartile Range); unit: bleeding episodes per year
Arm/Group | Arm B: Nonacog Beta Pegol (Prophylaxis)
Number analyzed (Participants) | 15
bleeding episodes per year | 3.12 [0.00 to 4.23]

3. Secondary Outcome: Consumption of Nonacog Beta Pegol for Treatment of Bleeding Episodes
Description: The mean number of injections of N9-GP used for treatment of a bleed from start to stop of a bleed was reported and it was measured in international units per kilogram per bleed (IU/kg/bleed).
Time Frame: From start of treatment (week 0) until end of treatment (up to week 50)
Population: Results were based on the FAS which included all participants exposed to N9-GP in this trial.
Measure: Mean (Standard Deviation); unit: IU/kg per bleed
Units Other Than Participants: Bleeding Episodes
Arm/Group | Arm A: Nonacog Beta Pegol (On-demand) | Arm A: Nonacog Beta Pegol (Prophylaxis) | Arm B: Nonacog Beta Pegol (Prophylaxis)
Number analyzed (Participants) | 15 | 14 | 15
Number analyzed (Bleeding Episodes) | 215 | 4 | 43
IU/kg per bleed | 42.4 (1.1) | 41.9 (0.5) | 41.6 (0.4)

4. Secondary Outcome: Consumption of Nonacog Beta Pegol for Prophylaxis (PPX) Treatment (Arm B Only)
Description: The mean consumption of N9-GP for prophylaxis per year per participant was reported and it was measured in international units per kilogram per year (IU/kg/year).
Time Frame: From start of treatment (week 0) until end of treatment (week 50)
Population: Results were based on the FAS which included all participants exposed to N9-GP in this trial.
Measure: Mean (Standard Deviation); unit: IU/kg per year
Arm/Group | Arm B: Nonacog Beta Pegol (Prophylaxis)
Number analyzed (Participants) | 15
IU/kg per year | 2212.3 (26.0)

5. Secondary Outcome: FIX Trough Levels During Prophylaxis (PPX) Treatment (Arm B Only)
Description: Trough levels of FVIII was reported for all participants who received prophylaxis treatment. Chromogenic assay was performed with N9-GP product specific standard (PSS) as a calibrator. The analysis is based on a mixed model on the log transformed plasma FVIII activity with age group as fixed effect and participants as a random effect. The mean trough is presented back-transformed to the natural scale. The estimated mean/average steady state trough level of FVIII over time (all visits from start of treatment (week 0) until end of treatment) was presented. Data is reported for specific treatment in which participants were a part of at any time from week 0 to end of the treatment (EOT) Week 50, not at specific time points assessed from week 0 to EOT.
Time Frame: From start of treatment (week 0) until end of treatment (week 50)
Population: Results were based on the FAS which included all participants exposed to N9-GP in this trial.
Measure: Mean (95% Confidence Interval); unit: International unit per milliliter(IU/mL)
Arm/Group | Arm B: Nonacog Beta Pegol (Prophylaxis)
Number analyzed (Participants) | 15
International unit per milliliter(IU/mL) | 0.298 [0.260 to 0.341]

6. Secondary Outcome: Number of Participants With Inhibitory Antibodies Against FIX Defined as Titre ≥0.6 Bethesda Units (BU)
Description: Number of participants who developed inhibitory antibodies (IA) against FVIII was presented. A participant was said to have FVIII-inhibitors if two consecutive tests, preferably within 2 weeks, were positive (greater than or equal to (≥) 0.6 bethesda unit (BU)). For the calculation of the inhibitor rate the numerator was included for all participants with neutralising antibodies while the denominator was included for all participants with a minimum of 50 exposures plus any participants with less than 50 exposures but with neutralising inhibitor.
Time Frame: From start of treatment (week 0) until end of treatment (week 50)
Population: Results were based on the FAS which included all participants exposed to N9-GP in this trial.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Nonacog Beta Pegol (On-demand) | Arm A: Nonacog Beta Pegol (Prophylaxis) | Arm B: Nonacog Beta Pegol (Prophylaxis)
Number analyzed (Participants) | 15 | 14 | 15
Participants | 0 | 0 | 0

7. Secondary Outcome: Number of Adverse Events (AEs)
Description: An adverse event (AE) was defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom or disease temporally associated with the use of a product, whether or not considered related to the product. All presented AEs are treatment-emergent. A treatment-emergent adverse event was defined as an event with onset after first N9-GP administration.
Time Frame: From start of treatment (week 0) until end of treatment (week 50)
Population: Results were based on the SAS which included all participants exposed to N9-GP in this trial.
Measure: Number; unit: Events
Arm/Group | Arm A: Nonacog Beta Pegol (On-demand) | Arm A: Nonacog Beta Pegol (Prophylaxis) | Arm B: Nonacog Beta Pegol (Prophylaxis)
Number analyzed (Participants) | 15 | 14 | 15
Events | 29 | 6 | 29

8. Secondary Outcome: Number of Serious Adverse Events (SAEs)
Description: A serious adverse event (SAE) is defined as any untoward medical occurrence that at any dose results in death, or is life-threatening, or requires inpatient hospitalization or causes prolongation of existing hospitalization results in persistent or significant disability/incapacity, or may have caused a congenital anomaly/birth defect, or requires intervention to prevent permanent impairment or damage. All presented SAEs are treatment-emergent (any serious adverse events which occurred after trial product administration).
Time Frame: From start of treatment (week 0) until end of treatment (week 50)
Population: Results were based on the SAS which included all participants exposed to N9-GP in this trial.
Measure: Number; unit: Events
Arm/Group | Arm A: Nonacog Beta Pegol (On-demand) | Arm A: Nonacog Beta Pegol (Prophylaxis) | Arm B: Nonacog Beta Pegol (Prophylaxis)
Number analyzed (Participants) | 15 | 14 | 15
Events | 1 | 0 | 0

9. Secondary Outcome: Incremental Recovery (IR) (Arm B Only)
Description: The incremental recovery was calculated by subtracting the FVIII activity (IU/mL) measured in plasma at time 0 from that measured at time 30 min after dosing and dividing this difference by the dose injected at time 0 expressed as international units per kilogram (IU/kg) body weight. FVIII activity was measured with a chromogenic assay.
Time Frame: Single-dose: 30±10 minutes post injection at week 0, Steady-state: 30±10 minutes post injection at week 12
Population: The Pharmacokinetic (PK) analysis set included sub-set of subjects from FAS who were included for PK assessments. Number analysed = Number of participants with available data for specific timepoints.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: (IU/mL)/(IU/kg)
Arm/Group | Arm B: Nonacog Beta Pegol (Prophylaxis)
Number analyzed (Participants) | 15
(IU/mL)/(IU/kg)
  Week 0: number analyzed (Participants) | 14
  Week 0 | 0.0182 (18.9550)
  Week 12 | 0.0192 (17.2668)

10. Secondary Outcome: Terminal Half-life (t½) (Arm B Only)
Description: Terminal half life was calculated as ln(2)/λz; where λz is the terminal elimination rate constant. The terminal elimination rate constant was estimated using linear regression on the terminal part of the log (activity) versus time profile.
Time Frame: Single-dose: 30±10 minutes post injection at week 0, Steady-state: 30±10 minutes post injection at week 12
Population: The PK analysis set included sub-set of participants from FAS who were included for PK assessments. Here, Number analysed (n) = Number of participants with available data for specific timepoints.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour
Arm/Group | Arm B: Nonacog Beta Pegol (Prophylaxis)
Number analyzed (Participants) | 15
hour
  Week 0: number analyzed (Participants) | 13
  Week 0 | 90.868 (13.535)
  Week 12 | 90.738 (21.581)

11. Secondary Outcome: Clearance (CL) (Arm B Only)
Description: Clearance (CL) of drug after intravenous administration was reported. Clearance was calculated using the formula CL= Dose / AUC(0-inf) for single dose and CL= Dose / AUC(0-96) h for steady state.
Time Frame: Single-dose: 0-168 hours post injection at week 0, Steady-state: 0-168 hours post injection at week 12
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milliliters per hour per kilogram
Arm/Group | Arm B: Nonacog Beta Pegol (Prophylaxis)
Number analyzed (Participants) | 15
milliliters per hour per kilogram
  Week 0: number analyzed (Participants) | 13
  Week 0 | 0.536 (22.143)
  Week 12 | 0.487 (26.552)

12. Secondary Outcome: Area Under the Curve (AUC) (Arm B Only)
Description: Area under the plasma activity versus time profile from time zero to 168 hours (AUC0-168h) was measured.
Time Frame: Single-dose: 0-168 hours post injection at week 0, Steady-state: 0-168 hours post injection at week 12
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours*international units per milliliter
Arm/Group | Arm B: Nonacog Beta Pegol (Prophylaxis)
Number analyzed (Participants) | 15
hours*international units per milliliter
  Week 0: number analyzed (Participants) | 14
  Week 0 | 51.856 (30.134)
  Week 12 | 92.914 (21.725)

ADVERSE EVENTS:
Time Frame: From start of treatment (Week 0) until end of trial (Week 54)
Description: All presented AEs are treatment-emergent adverse events. A TEAE was defined as an event with onset after first N9-GP administration. Results were based on the SAS which included all participants exposed to N9-GP in this trial.
Arm/Group | Arm A: Nonacog Beta Pegol (On-demand) | Arm A: Nonacog Beta Pegol (Prophylaxis) | Arm B: Nonacog Beta Pegol (Prophylaxis)
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/14 | 0/15
Serious Adverse Events (participants affected / at risk) | 1/15 | 0/14 | 0/15
Other Adverse Events (participants affected / at risk) | 12/15 | 4/14 | 14/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: Nonacog Beta Pegol (On-demand) (N=15) | Arm A: Nonacog Beta Pegol (Prophylaxis) (N=14) | Arm B: Nonacog Beta Pegol (Prophylaxis) (N=15)
Haematoma infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: Nonacog Beta Pegol (On-demand) (N=15) | Arm A: Nonacog Beta Pegol (Prophylaxis) (N=14) | Arm B: Nonacog Beta Pegol (Prophylaxis) (N=15)
Acne (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Atrioventricular block (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Blood fibrinogen decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood fibrinogen increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
C-reactive protein increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0) | 6 (6)
Chest discomfort (General disorders) | 0 (0) | 1 (1) | 0 (0)
Coronavirus infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (3)
Fibrin D dimer increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Fibrinogen degradation products increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Haemophilic arthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2)
Hypoproteinaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 1 (1) | 0 (0) | 0 (0)
Lymphadenitis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Neuritis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Periodontitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Phlebitis superficial (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Procalcitonin increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 2 (2) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Synovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Trichiasis (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 4 (5)
Weight increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
White blood cell count increased (Investigations) | 1 (2) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At the end of the trial, one or more scientific publications may be prepared collaboratively by the investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for up to 60 days to protect intellectual property.

DOCUMENTS (2):
  • Study Protocol (2021-09-22): https://cdn.clinicaltrials.gov/large-docs/17/NCT05365217/Prot_000.pdf
  • Statistical Analysis Plan (2021-02-03): https://cdn.clinicaltrials.gov/large-docs/17/NCT05365217/SAP_001.pdf